## **INFORMATION**

A study on intensive rehabilitation of language and speech after brain injury



At Karolinska Institutet, we are conducting a study on how intensive training can affect language and speech ability after a stroke.

The study is conducted at Hedla Intensive Rehab.



The purpose of the study is to develop better treatments for people who have problems with their language or speech after a brain injury.

If you participate in the study, you agree that we use your test results and brain scans in research.









We save your test results, but without your name. We also save information about your age, sex, diagnosis and where in the brain your injury has affected you.



The material is coded and can't be connected to you. All personal data is protected by confidentiality and the EU Data Protection Act (GDPR).

- It is **voluntary** to participate in the study.
- You can end your participation at any time without affecting your continued rehabilitation.
- You do not receive any compensation for participating in the study.



 According to the EU Data Protection Act (GDPR), you have the right to access information about you, and have it revised, corrected or deleted.







If you agree to be included in the study, your rehab will consist of at least **3 hours of speech training** per day for ten days of the program. Other planned training is not affected.



Testing of speech, language and quality of life takes place on three occasions, the last testing is done in your hometown. Testing of motor functions and cognition takes place immediately before and after intensive speech training.



You will do magnetic resonance imaging (MRI) of the brain at the University of Malaga before and after completing language and speech training.







- A doctor examine you to rule out risk factors such as pacemakers or pieces of metal implanted in your body before the procedure.
- The examination has no known risks, but it can be perceived as unpleasant to lie still on a bunk in the narrow space in the magnetic camera.
- The examination takes about 40 60 minutes.

Responsible for the research and personal data controller is Karolinska Institutet.

If you have questions about how the information is processed, you can contact: KI's data protection representative (<u>dataskyddsombud@ki.se</u>) or Datainspektionen (datainspektionen.se)

## Principal researcher / contact person:

Ellika Schalling, Associate Professor, Speech Language Pathologist, Division of Speech and Language Pathology, Department of Clinical Science, Intervention and Technology, Karolinska Institutet,

Phone: 08-5248 8912, e-mail: ellika.schalling@ki.se

Participating researcher and responsible for conducting assessments:

Marika Schütz, Speech Language Pathologist, doctoral student at Karolinska Institutet. Phone: 0737570430, e-mail: marika.schutz@ki.se

Consent to participate in the study:

## Evaluation of effects regarding speech, language, communication and quality of life after two weeks of intensive speech therapy treatment

I have received oral, image-supported and written information about the study and have had the opportunity to ask questions. I may keep the written image-supported information. I have understood what the research study entails and I agree to participate in the study and to have my personal data handled in the way that appears from the information I have received.

## I want to be part of this study



Principal researcher / contact person: Ellika Schalling, Associate Professor, Speech Language Pathologist, Unit of Speech Therapy, Department of Clinical Science, Intervention and Technology, Karolinska Institutet,

Phone: 08-5248 8912, e-mail: ellika.schalling@ki.se

Consent obtained from

Participating researchers and responsible for conducting surveys: Marika Schütz, Speech Language Pathologist, doctoral student at Karolinska Institutet.

Phone: 0737570430, e-mail: marika.schutz@ki.se